CLINICAL TRIAL: NCT05851469
Title: An Explorative, Non-randomized, Open-label, In-clinic Study, Investigating the Performance of a Novel Non-invasive Glucose Monitoring Device Using a New Guided Calibration Model
Brief Title: Study of a Non-invasive Glucose Measuring Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RSP Systems A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: RSP-26
Record Dates: First submitted 2023-03-31; First posted 2023-05-09 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus
Keywords: Non-invasive; Blood sugar; Raman spectroscopy
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RSP-26-01 (Experimental)
  Interventions: Device: Prototype 0.5
- RSP-26-02 (Experimental)
  Interventions: Device: Prototype 0.5

INTERVENTIONS:
Device: Prototype 0.5 — Investigational Medical Device collecting Raman data from tissue

SUMMARY:
This explorative clinical investigation has been launched to collect spectral Raman data paired with validated glucose reference values in persons with diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject ≥18 years.
2. Subject with type 2 diabetes.
3. Signed informed consent form (ICF).

Exclusion Criteria:

1. Individual treated with intensified insulin treatment.
2. Sodium, Potassium. Creatinine, eGFR, and ALAT (more than three times the upper limit of normal range).
3. Clinically relevant anaemia or thrombocytopenia.
4. Infection with hepatitis B, C or HIV (if subject participates in subprotocol 1).
5. Intake of anticoagulant medication (with the exception of acetylsalicylic acid, ASS 100).
6. For female subjects: Pregnancy or breastfeeding or lack of a negative pregnancy test (except in case of menopause, sterilization, or hysterectomy).
7. Subjects not able to understand and read local language.
8. Cognitive impairment, or in investigator's opinion, subject is not able to follow instructions provided and as specified in the clinical investigation plan (CIP).
9. Subject not able to hold hand/arm steady (including tremors and Parkinson's Disease).
10. Skin changes, tattoos, or diseases on right thenar (measurement site).
11. Reduced circulation in right hand evaluated by Allen's test.
12. Known allergy to medical grade alcohol.
13. Haemodialysis.
14. Topical administration of glucocorticoids at the right hand for the past 7 days or during the study period.
15. Any disorder, which in the investigator's opinion, might jeopardise subject's safety or compliance with the CIP.
16. Any incapacity or general condition that, in the opinion of the investigator, prevents adequate compliance with the study procedures, e.g., mental, or visual incapacity, language barriers, alcohol or drug abuse.
17. Dependency from the sponsor or the clinical investigator (e.g., co-workers of the sponsor, the study site, and/ or their families).
18. Subjects currently participating in another study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
Clinical performance | 2 days
  Repeated measurements of blood sugar, to cover the diurnal variation, with the non-invasive examination device, and compare the result with blood drawn capillary and venous

SECONDARY OUTCOMES:
Adverse events | 4 days
  Frequency of adverse reactions related and non-related to the investigational device

CONTACTS AND LOCATIONS:
Locations (1):
- Institut für Diabetes-Technologie, Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm, Ulm, Germany